CLINICAL TRIAL: NCT02768519
Title: A Phase 1, Randomised, Placebo-controlled, Double-blind, Cross-over Study to Evaluate Systemic Bioavailability of Oral OTS167 Under Fed and Fasting Conditions in Healthy Adult Subjects
Brief Title: Study to Evaluate Systemic Bioavailability of Oral OTS167 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OTS167-FR03
Record Dates: First submitted 2016-04-13; First posted 2016-05-11 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- OTS167IV (Experimental): Cohort 1: 0.5 mg, Cohort 2: 1.0 mg, and Cohort 3: 2.0 mg without food on Period 1 Day 1 and with food on Day 1 Period 2.
  Interventions: Drug: OTS167IV
- Placebo (Placebo Comparator): Cherry syrup
  Interventions: Other: Cherry syrup

INTERVENTIONS:
Drug: OTS167IV — diluted to final concentration with cherry syrup
  Arms: OTS167IV
Other: Cherry syrup
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the indicative bioavailability of a single oral dose of OTS167, and to evaluate the effects of food on OTS167 pharmacokinetics (PK) after oral dosing.

Eleven male and female healthy participants aged 45 years and over will be entered into this phase 1, single-centre, double-blind, randomised, cross-over study. The trial is designed to evaluate the bioavailability of OTS167, and the effects of food on pharmacokinetics (PK) of OTS167 when administered by the oral route. Correlative studies include evaluation of safety endpoints and examinations, and adverse events. This study involves 3 cohorts to evaluate the safety and tolerability of oral dosing from lower dose.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following criteria to be eligible for participation in the study:

1. Males or females aged 45 years or over.
2. Female participants of non-childbearing potential, meeting at least one of the following criteria:

   * Amenorrhoeal for 12 months (menopause confirmed by Follicular Stimulating Hormone (FSH) and Luteinising Hormone (LH) levels as defined by the established reference ranges), or
   * Surgically sterile (e.g. hysterectomy, oophorectomy, tubal ligation) for at least the past 3 month.
3. Able to communicate with site personnel and to understand and voluntarily sign the Informed Consent Form (ICF).
4. Able and willing to comply with the protocol, including availability for all scheduled study visits.
5. Body mass index (BMI) 18 kg/m2 to 30 kg/m2 (inclusive)
6. No clinically significant abnormalities as determined by medical history, physical examination, blood chemistry, hematology, urinalysis, and 12-lead electrocardiogram (ECGs).
7. If male, agrees to use a medically acceptable method of contraception from Screening until 7 days after administration of the last dose of study drug. Medically acceptable methods of contraception include the following: abstinence; medically approved hormonal methods; condom; diaphragm; and intrauterine device. This requirement may be waived if the Principal Investigator or delegate is satisfied that the participant or partner is sterile (i.e., if female has undergone a hysterectomy, or has undergone a tubal ligation at least 3 months prior to Screening, or is postmenopausal [no menstrual period for at least 12 months prior to Screening]; if male, has undergone vasectomy at least 6 months prior to Screening). Male participants agree not to donate sperm for at least 90 days [3 months] after administration of the last dose of study drug.
8. Agree to avoid drinking alcohol within 72 hours prior to check-in to the clinical facility.
9. Adequate venous access in the left and right arm to allow collection of a number of blood samples.

Exclusion Criteria: Participants meeting any of the following criteria are ineligible for participation in the study.

1. Evidence or history of clinical significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic diseases
2. Orthostatic blood pressure changes (>15mmHg) or symptoms, or presence of uncontrolled hypertension (SBP >160 mmHg or diastolic >95 mmHg) at screening, admission (Day -1) or pre-dose (Day 1).
3. Greater than 2 standard drinks per day, on average, for men and women, or any history of drug or alcohol addiction or abuse within the last 5 years.
4. History of allergic, anaphylaxis or hypersensitivity to OTS167 or excipients or contents of Humco ™ cherry syrup.
5. Female participants who are currently lactating.
6. Donated either blood or plasma (e.g., plasmapheresis) within 6 weeks prior to dosing in Period 1. All participants must be advised not to donate either blood or plasma for at least 6 weeks after completing the study.
7. Use of prescription medications (with the exception of contraceptives), over-the-counter medications (with the exception of paracetamol [< 2 gm/day] or single-dose daily multivitamins), or herbal medications or products containing herbal extracts within 14 days prior to the first dose.
8. Positive results on illicit drug test or alcohol breath test at screening or at admission.
9. Positive screening test for HIV antibodies, Hepatitis B surface antigen or Hepatitis C antibody.
10. Use of any investigational drug within the last 30 days or within a period of 5 times the drug's half-life, whichever is longer, or current participation in any investigational protocol.
11. Participants who, in the opinion of the Principal Investigator or delegate, should not participate in the study or are not capable of following the study schedule for any reason.
12. Either QTcF >450 or HR <40 or >100 at screening, admission (Day-1) or pre-dose (Day 1). Test may be repeated at discretion of investigator to obtain average in order to confirm eligibility.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety: Participants to be monitored throughout the treatment and follow-up period for occurrence of adverse events (AEs) (acute, delayed, and/or cumulative), as well as for changes in clinical status, vital signs, and laboratory data. | 7 days after final study drug administration.
  Safety assessments include concomitant medication survey, adverse events, temperature, pulse and respiratory rate, blood pressure, physical examination, hematologic parameters, serum chemistries, coagulation parameters, urinalyses, and 12-Lead ECG and cardiac telemetry.
Maximum Plasma Concentration (Cmax) | 24 hours after final study drug administration.
Time of Maximum concentration (Tmax) | 24 hours after final study drug administration.
Area Under the Curve (AUC) | 24 hours after final study drug administration.
Half life (T1/2) | 24 hours after final study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Principal Investigator — CMAX (A division of IDT Australia Ltd)
Locations (1):
- CMAX, Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided